CLINICAL TRIAL: NCT02291198
Title: Open Label, Prospective, Cross-Sectional Clinical Performance Study of the in Vitro Diagnostic Device NK Vue Kit: Measurement of Natural Killer Cell Activity in Whole Blood in Subjects Being Screened for Colorectal Cancer Using Colonoscopy
Brief Title: Measurement of NK Cell Activity in Whole Blood in Subjects Being Screened for Colorectal Cancer Using Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ATGen Canada Inc (Industry)
Collaborators: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ATG-001
Record Dates: First submitted 2014-11-10; First posted 2014-11-14 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Natural Killer Cell Cytokine Production
Keywords: colorectal cancer; natural killer cell activity; screening; NK cells
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NK Vue: NK cell activity in stimulated whole blood — One mL of blood is collected from each subject, on the day of colonoscopy, using NK Vue Promoca Tubes blood collection tubes containing a proprietary stimulating cytokine. After incubation, NK cell activity is measured in the collected plasma using an ELISA.

SUMMARY:
This study will look at measuring the activity of natural killer (NK) cells using the in vitro diagnostic device NK Vue in subjects being screened for colorectal cancer using colonoscopy. The NK Vue diagnostic test for natural killer cell activity uses the principle of stimulation of whole blood with a proprietary cytokine followed by the quantitative detection of interferon gamma using an immunoassay. NK Vue is intended to be used for the monitoring of the immune status of individuals. Measurement of NK cell activity could be a useful tool for assessing changes in immunosurveillance in patients with conditions or diseases where NK cell activity has been shown to be reduced, such as colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing colonoscopy at the hospital
* Subjects who have adequately prepared for their colonoscopies as per their doctor's directions
* Subjects whose colonoscopy preparation has been deemed to be excellent or sufficient during the colonoscopy procedure
* Subjects who provide informed consent to participate in the trial
* Subjects >40 years of age

Exclusion Criteria:

* Lack of understanding and/or participation due to illiteracy
* History of Active viral or bacterial infection
* History of prescription use of immunosuppressive drugs within the last six months
* History of anticancer treatments including surgery or chemotherapy
* History of autoimmune disorders (rheumatoid arthritis, multiple sclerosis, systemic lupus erythematosus, inflammatory bowel disease including Crohn's disease, Type I diabetes, Guillain-Barré syndrome)
* Known HIV, Hepatitis B, or Hepatitis C infection
* Currently participating (or participated within the previous 120 days) in an investigational therapeutic or device study
* Female who is pregnant, nursing, or of child-bearing potential while not practicing effective contraceptive methods.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1081 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
NK cell activity | Blood drawn for NK cell activity on day of colonoscopy
  Measurement of NK cell activity in subjects with cancer-negative colonoscopies versus those with pathologically confirmed colorectal cancer.
  Correlation of NK cell activity with polyp size, with type of adenomatous polyp and with cancer stage; measurement of the sensitivity and specificity of NK Vue; determination of the positive predictive value of NK Vue alone or in combination with the fecal immunochemical test in those subjects positive for adenomatous polyps or cancer; determination of the impact of performing both NK Vue and the fecal test on the sensitivity of the fecal test.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Jobin, MD, FRCP, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Hopital Maisonneuve-Rosemont, Montreal, Quebec, Canada

REFERENCES:
- [Background] Lee SB, Cha J, Kim IK, Yoon JC, Lee HJ, Park SW, Cho S, Youn DY, Lee H, Lee CH, Lee JM, Lee KY, Kim J. A high-throughput assay of NK cell activity in whole blood and its clinical application. Biochem Biophys Res Commun. 2014 Mar 14;445(3):584-90. doi: 10.1016/j.bbrc.2014.02.040. Epub 2014 Feb 18. PMID 24561245
- [Background] Koo KC, Shim DH, Yang CM, Lee SB, Kim SM, Shin TY, Kim KH, Yoon HG, Rha KH, Lee JM, Hong SJ. Reduction of the CD16(-)CD56bright NK cell subset precedes NK cell dysfunction in prostate cancer. PLoS One. 2013 Nov 4;8(11):e78049. doi: 10.1371/journal.pone.0078049. eCollection 2013. PMID 24223759
- [Background] Kim JC, Choi J, Lee SJ, Lee YA, Jeon YM, Kang YW, Lee JK. Evaluation of cytolytic activity and phenotypic changes of circulating blood immune cells in patients with colorectal cancer by a simple preparation of peripheral blood mononuclear cells. J Korean Surg Soc. 2013 Nov;85(5):230-5. doi: 10.4174/jkss.2013.85.5.230. Epub 2013 Oct 25. PMID 24266014
- [Background] Furue H, Matsuo K, Kumimoto H, Hiraki A, Suzuki T, Yatabe Y, Komori K, Kanemitsu Y, Hirai T, Kato T, Ueda M, Ishizaki K, Tajima K. Decreased risk of colorectal cancer with the high natural killer cell activity NKG2D genotype in Japanese. Carcinogenesis. 2008 Feb;29(2):316-20. doi: 10.1093/carcin/bgm260. Epub 2008 Jan 3. PMID 18174257
- [Background] Hayashi T, Imai K, Morishita Y, Hayashi I, Kusunoki Y, Nakachi K. Identification of the NKG2D haplotypes associated with natural cytotoxic activity of peripheral blood lymphocytes and cancer immunosurveillance. Cancer Res. 2006 Jan 1;66(1):563-70. doi: 10.1158/0008-5472.CAN-05-2776. PMID 16397273
- [Background] Imai K, Matsuyama S, Miyake S, Suga K, Nakachi K. Natural cytotoxic activity of peripheral-blood lymphocytes and cancer incidence: an 11-year follow-up study of a general population. Lancet. 2000 Nov 25;356(9244):1795-9. doi: 10.1016/S0140-6736(00)03231-1. PMID 11117911
- [Result] Jobin G, Rodriguez-Suarez R, Betito K. Association Between Natural Killer Cell Activity and Colorectal Cancer in High-Risk Subjects Undergoing Colonoscopy. Gastroenterology. 2017 Oct;153(4):980-987. doi: 10.1053/j.gastro.2017.06.009. Epub 2017 Jun 15. PMID 28625834